CLINICAL TRIAL: NCT05960682
Title: French Translation and Validation of the Brief Index of Sexual Functioning for Men
Acronym: FraQBISFM
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0260
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sexual Dysfunction Male
Keywords: Sexual Dysfunction Male
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Men will complete the French version of the Brief Index of Sexual Functioning for Men paper questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will complete the French version of the Brief Index of Sexual Functioning for Men (BISFM) paper questionnaire. The BISFM is a self-administered questionnaire. It has 22 questions, grouped into 7 domains allowing a qualitative and quantitative evaluation of the sexual experience: D1 (desire), D2 (excitement), D3 (frequency of activity), D4 (receptivity), D5 (pleasure, orgasm ), D6 (relationship satisfaction), D7 (problems affecting sexuality).

SUMMARY:
Sexual dysfunction consists of a disorder of the sexual response, either in terms of desire, or in terms of vasocongestion, or in terms of orgasmic response, or in more than one phase of this response :

Sexual dysfunctions are today described by the Diagnostic and Statistical Manual (DSM) V as:

* Disorders of sexual desire or decreased libido
* Sexual arousal disorder
* Delayed or absent orgasmic disorder
* Sexual disorder with pain Moreover, sexual dysfunctions are not without consequences on the life of a couple. The origins of these dysfunctions are multiple, but the result is most of the time the same: fear of failure, feeling of incompetence, anxiety, frustration or misunderstanding.

To date, the scientific community benefits from a few self-administered questionnaires to measure the impact of certain dysfunctions. None takes into account all the dimensions of male sexuality. In Italy, the Brief Index of Sexual Functioning for Men is used. This questionnaire contains 22 items, grouped into 7 areas exploring all of male sexuality: desire, arousal, frequency of activity, receptivity, pleasure/orgasm, relationship satisfaction, problem affecting sexuality. This questionnaire is not currently validated in French, whereas the Brief Index of Sexual Functioning for Women is validated.

DETAILED DESCRIPTION:
In this context, the Andrology Committee of the French Association of Urology wishes to create a pilot study with French patients presenting sexual dysfunctions with the aim of validating the questionnaire in French. Patient responses to each item will:

* to determine if the formulation of the items is understandable by all, or if this is not the case
* to identify the difficulties it can cause, and their causes. Patients treated for sexual dysfunction will be informed of the possibility of answering a questionnaire and that their data will be recorded for the purpose of studying practices and analyzing the results in an anonymous setting, and confidential via the delivery of the information leaflet dedicated to the study. They will have the opportunity to signify their refusal to participate without risk of modification of the coverage.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with sexual dysfunction

Exclusion Criteria:

* Patient refusing to participate
* Patient with difficulties in understanding the French language.
* Protected persons referred to in Articles L.1121-6 to L.1121-8 of the Public Health Code

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Questionnary oly for men
Study Population: Adult mens treated for sexual dysfunction at the Toulouse University Hospital
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Response rate to the paper questionnaire | Day 1
  Answer two sub-questions a) and b) after each item of the scale. These answers will allow to determine if the formulation of the items is understandable by all, or if this is not the case, to identify the difficulties it can cause, and their causes.

CONTACTS AND LOCATIONS:
Overall Officials: Eric HUYGHE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Hospital, Toulouse, France